CLINICAL TRIAL: NCT02131688
Title: Phase I Dose Escalation Study of Mitoxantrone Hydrochloride Liposome Injection in Patients With Malignant Lymphoma
Brief Title: Phase I Study of Mitoxantrone Hydrochloride Liposome Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HE14Ⅰ
Record Dates: First submitted 2014-05-04; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-03

CONDITIONS: Malignant Lymphoma
Keywords: safety;malignant lymphoma;
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome (Experimental)
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose,the safety and effectiveness of Mitoxantrone Hydrochloride Liposome Injection.

DETAILED DESCRIPTION:
The trial of the dose escalation method is from 18mg/m2 until the maximum tolerated dose and every 3 patient is a dose group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must compliance with the requirements and restrictions listed in the consent form
* Patients with Pathology and / or cytologically proven malignant lymphoma
* Patients must be 18-70 years old ,both male and female
* Failure of standard chemotherapy
* Patients have no better choice and may be benefit from the use of anthracyclines
* Patients with Eastern Cooperative Oncology Group (ECOG)Performance Status of 0-2
* Objective tumor from the last chemotherapy, biological therapy or other experimental interval treatment least 4 weeks
* Expected survival time ≥ 3 months
* Patients agreed to take effective contraceptive measures during the trial
* Blood routine, liver and kidney function, cardiac function examination in accordance with the following requirements.

Exclusion Criteria:

* Pregnancy and breast-feeding women
* Multiple sclerosis
* Patients that have histories of ischemic heart disease and heart congestive,arrhythmia that need to be a treatment and significant valvular disease
* Patients with heart disease induced by anthracycline
* Patients requiring other antineoplastic treatment
* Patients with temperature above 38 degrees or active infection that may effects in clinical tests
* Patients are allergic to anthracycline and liposomal drugs
* Patients are allergic to eggs,egg products,soybean and soybean products
* Patients with uncontrolled primary or metastatic brain tumorsMultiple sclerosis
* Patients that have histories of ischemic heart disease and heart congestive,arrhythmia that need to be a treatment and significant valvular disease
* Patients with heart disease induced by anthracycline
* Patients requiring other antineoplastic treatment
* Patients with temperature above 38 degrees or active infection that may effects in clinical tests
* Patients are allergic to anthracycline and liposomal drugs
* Patients are allergic to eggs,egg products,soybean and soybean products
* Patients with uncontrolled primary or metastatic brain tumors
* Total amount of Doxorubicin(or Pirarubicin)≥360mg/m2,Epirubicin ≥600mg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Mitoxantrone Hydrochloride Liposome Injection | 4 months

SECONDARY OUTCOMES:
Objective Response Rate | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Ph.D, Principal Investigator — Cancer Hospital ,Chinese Academy of Mddical Sciences
Locations (1):
- Cancer Hospital ,Chinese Academy of Mddical Sciences, Beijing, China